CLINICAL TRIAL: NCT03738358
Title: A 12-week, Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Study to Evaluate the Efficacy and Safety of Trehalose in Patients With Fatty Liver Disease
Brief Title: Clinical Study of 12-week Trehalose Intake in Patients With Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Ryul Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-02-015
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Non-alcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Trehalose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trehalose (Experimental)
  Interventions: Dietary Supplement: Trehalose
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Trehalose — 80 mL pouch/day for 12 weeks, containing trehalose 5 g, water 74.92 g and scent additive 0.08 g
  Arms: Trehalose
Other: Placebo — 80 mL pouch/day for 12 weeks, containing water 79.92 g and scent additive 0.08 g
  Arms: Placebo

SUMMARY:
This clinical study will be conducted to evaluate the efficacy and safety of trehalose in patients with fatty liver disease. After 12-week intake, subjects will be checked up fat content in liver using CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19-year-old and 79-year-old
* Weight (≥50kg)
* Is diagnosed as fatty liver on ultrasonography within 24 weeks from screening day
* Has willingness and ability to participate whole clinical study period
* Willing to give informed consent form

Exclusion Criteria:

* Patient with alcoholic fatty liver
* Patient with inflammatory bowel disease
* Is required treatment for like liver, kidney, digestive system, circulatory system, respiratory system, endocrine system(except diabetes), musculoskeletal, neuropsychiatry, or hemato-oncology etc., which is able to effect on clinical study
* Has any medical history with virus or toxic hepatitis
* Has any medical history of gastrointestinal surgery (except simple appendectomy & repair of hernia)
* Has medical history of malignant tumor (except non-melanoma skin cancer) within the last 5 years from the screening day
* Took any drugs (UDCA, silymarin, omega-3, fenofibrate etc.) which is decided as unsuitable drug for combined-dose by investigator
* Over 4 times of maximum reference range of ALT or AST
* Average drinking quantity per week > alcohol 140 g
* Pregnant or nursing women
* Is currently participating into another clinical study
* Being made a decision from investigator as unsuitable to participate this study

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content scanned by CT | Screening (baseline) and 12 weeks
  Trehalose group and placebo comparator group are scanned by CT to compare the difference of liver fat content

SECONDARY OUTCOMES:
Change in ALT and AST | 0 (baseline) and 12 weeks
  Change from baseline of ALT and AST, the trend of change in blood, the proportion of subjects with normal ALT and AST level
Change in homeostatic model assessment-insulin resistance (HOMA-IR) | Screening (baseline) and 12 weeks
  Change from baseline of HOMA-IR, the trend of change in blood, the proportion of subjects with normal HOMA-IR level
Change in total cholesterol, LDL, HDL, triglyceride (TG) and free fatty acid | 0 (baseline), 6 and 12 weeks
  the trend of change in blood
Change in BMI | 0 (baseline), 6 and 12 weeks
  BMI among subjects is measured by physical examination
Change in visceral fat and subcutaneous fat levels | 0 week and 12 weeks
  Both visceral fat and subcutaneous fat levels are anlayzed by CT scan.
Adverse event (AE) | 0 week, 6 weeks, and 12 weeks
  Symptom and signs in subjects are monitored